CLINICAL TRIAL: NCT02531113
Title: A Phase 2, Multi-Center, Open-Label Induction Trial With Extension Period to Access Endoscopic Improvement and Changes in Intestinal and Serum Biomarkers in Patients With Moderately to Severely Active Crohn's Disease Receiving Oral RPC1063 as Induction Therapy
Brief Title: Efficacy and Safety Trial of RPC1063 for Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPC01-2201
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RPC1063 (Ozanimod) (Experimental)
  Interventions: Drug: RPC1063

INTERVENTIONS:
Drug: RPC1063
  Other Names: Ozanimod

SUMMARY:
The purpose is to determine whether RPC1063 is effective in the treatment of Crohn's disease.

DETAILED DESCRIPTION:
This open-label trial is composed of two periods: Induction and Extension. All eligible patients will be enrolled into the 12-Week Induction period and receive study medication. Patients who complete the Induction period may then be eligible to enter the 100-Week Extension period where they will continue to receive study medication.

ELIGIBILITY:
Key Inclusion Criteria:

* Crohn's disease (CD) confirmed by endoscopy and histology
* Active disease as evaluated by Crohn's Disease Activity Index Score and Simple Endoscopic Score for CD
* Inadequate response to aminosalicylates, corticosteroids, immunomodulators or biologic therapy

Key Exclusion Criteria:

* Diagnosis of ulcerative colitis or indeterminate colitis
* Known strictures/stenosis leading to symptoms of obstruction
* Current stoma or need for ileostomy or colostomy
* Clinically relevant cardiovascular conditions or other relevant diseases that could impact the implementation or interpretation of the trial, or put the patient at risk
* History of uveitis or known macular edema
* History of colonic dysplasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanthi Kollengode, MD, Study Director — Celgene Corporation
Locations (28):
- United States (13):
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Florida Center for Gastroenterology, Largo, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Atlanta Gastroenterology Specialists PC, Suwanee, Georgia
  - DM Clinical Research, Oak Lawn, Illinois
  - Gastroenterology Associates LLC, Baton Rouge, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Ehrhardt Clinical Research LLC, Belton, Missouri
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Gastro One, Germantown, Tennessee
  - San Antonio Gastroenterology, San Antonio, Texas
- LHSC Victoria Hospital, London, Ontario, Canada
- Hungary (2):
  - Szent Margit Korhaz, Budapest
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
- Poland (5):
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - GASTROMED Sp.zo.o., Lublin
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Centralny Szpital Kliniczny MSWIA, Warsaw
  - Nzoz Vivamed, Warsaw
- Ukraine (7):
  - Si Institute Of Gastroenterology Of Namsu Dept Of Stomach And Duodenum Diseases, Dnipropetrovsk
  - Kharkiv City Clinical Hospital 2, Kharkiv
  - Municipal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Kyiv CCH #18 Dept of Proctology O. O. Bogomolets NMU, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Vinnytsia Regional Clinical, Vinnytsia
  - CI City Hospital #1, Zaporizhia

REFERENCES:
- [Derived] Harris S, Feagan BG, Hanauer S, Vermeire S, Ghosh S, Yan J, Wu C, Hu Y, Maddux R, Wolf DC, D'Haens G. Ozanimod Differentially Impacts Circulating Lymphocyte Subsets in Patients with Moderately to Severely Active Crohn's Disease. Dig Dis Sci. 2024 Jun;69(6):2044-2054. doi: 10.1007/s10620-024-08391-z. Epub 2024 Apr 3. PMID 38568396
- [Derived] Feagan BG, Sandborn WJ, Danese S, Wolf DC, Liu WJ, Hua SY, Minton N, Olson A, D'Haens G. Ozanimod induction therapy for patients with moderate to severe Crohn's disease: a single-arm, phase 2, prospective observer-blinded endpoint study. Lancet Gastroenterol Hepatol. 2020 Sep;5(9):819-828. doi: 10.1016/S2468-1253(20)30188-6. Epub 2020 Jun 15. PMID 32553149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-nine adult participants were enrolled from 28 sites located in Europe and North America.
Pre-assignment Details: Eligible participants must have had a Crohn's Disease Activity Index (CDAI) score of 220 to 450 inclusive with an Simple Endoscopic Score for Crohn's Disease (SES-CD) score of ≥ 6 and an average daily stool score ≥ 4 points and/or an average daily abdominal pain score of ≥ 2 points.
Groups:
- Ozanimod Hydrochloride (HCl) 1 mg: Participants received ozanimod 1 mg capsules daily for the first 12 weeks of the induction period (an initial 7-day dose escalation regimen that consisted of 4 days of ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg) daily followed by 3 days of ozanimod HCl 0.5 mg (equivalent to ozanimod 0.46 mg) daily, with the final dose of ozanimod HCl 1 mg (equivalent to ozanimod 0.92 mg) daily dose reached on Day 8. Participants who completed the induction period had the opportunity at Week 12 to continue to receive ozanimod 1 mg capsules daily during the extension period up to an additional 148 weeks, provided that the investigator determined that the participant should continue. Participants in the extension period continued to receive ozanimod 1 mg capsules daily through Week 160. Participants who completed the Week 160 visit had the option to continue open-label ozanimod 1 mg capsules by immediately entering the open-label extension Phase 3 Crohn's Disease Study RPC01-3204 (NCT03467958).
Period: Induction Period: Week 0 to 12
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Started | 69
Completed (Completed = completed induction period and eligible to enter extension period.) | 58
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 3
Period: Extension Period: Week 12 up to Week 160
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Started | 52 (6 participants completed induction; did not advance to extension due to lack efficacy.)
Completed (Completed = Defined as participants who had 160 visit) | 14
Not Completed | 38
Not completed — Physician Decision | 2
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 19
Not completed — Withdrawal by Subject | 11
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat population included all enrolled participants who received at least one dose of investigational product (IP).
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 7
  Other | 1
  White | 60
Years Since Crohn's Disease Diagnosis [Mean (Standard Deviation); unit: Years] | 8.9 (8.53)
Crohn's Disease Activity Index (CDAI) Score at Baseline [Mean (Standard Deviation); unit: Units on a Scale] — The CDAI is a composite score that was used to measure the clinical activity of Crohn's disease. The CDAI used a questionnaire with responses scored numerically and weighted. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity.
  Units on a Scale | 322.8 (59.19)
Daily Stool Frequency (SF) at Baseline [Mean (Standard Deviation); unit: Stools/day] — SF = the average daily stool score = average of the number of liquid/soft stools for the available days in the 7-day window, using the most recent 7 days prior to the visit.
  Stools/day | 6.15 (2.792)
Daily Abdominal Pain Score at Baseline [Mean (Standard Deviation); unit: Units on a Scale] — The daily abdominal pain score was defined as the average of the abdominal pain level for the available days in the 7-day window, using the most recent 7 days prior to the visit date. Abdominal pain is scored on a scale 0-3.
  Units on a Scale | 2.05 (0.526)
Prior Corticosteroid Use [Count of Participants; unit: Participants]
  Prior Use of Corticosteroids | 62
  No Prior Use of Corticosteroids | 7
Simple Endoscopic Score for Crohn's Disease (SES-CD) at Baseline [Mean (Standard Deviation); unit: Units on a Scale] — The SES-CD assesses the degree of inflammation on the basis of 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 to 3 (worst). In the SES-CD, each of these 4 components were assessed in the five segments of the ileum and colon: ileum, right, transverse, left (descending and sigmoid), and rectum. The SES-CD is the sum of the individual scores of each of the components across the five segments, with higher scores indicating greater disease activity.
  Units on a Scale | 13.28 (6.584)
Prior Use of Immunomodulator [Count of Participants; unit: Participants]
  Prior Use of Immunomodulator | 38
  No Prior Use of Immunomodulator | 31
Fecal Calprotectin at Baseline [Mean (Standard Deviation); unit: μg/g] | 1158.17 (1231.267)
C-reactive Protein (mg/L) at Baseline [Mean (Standard Deviation); unit: (mg/L)] | 18.2 (25.36)
Disease Location [Count of Participants; unit: Participants]
  Ileum Only | 11
  Colon Only | 26
  Ileocolonic (Ileum and Colon) | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Simple Endoscopic Score for Crohn's Disease (SES-CD) (Paired Segments) From Baseline at Week 12 as Determined by a Blinded Central Reader.
Description: The simple endoscopy score (SES-CD) assesses the degree of inflammation. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components are scored on a scale of 0 to 3. In the SES-CD, each of these 4 components are assessed in the five segments of the ileum and colon: ileum, right, transverse, left (descending and sigmoid), and rectum. The SES-CD is the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores is 0 - 12 for each segment, and 0 - 56 for the overall SES-CD score, with larger scores indicating greater severity of disease.
Time Frame: Baseline to Week 12
Population: The intent to treat population = all enrolled participants who received at least one dose of ozanimod. For paired segment scores, any missing segment scores, were imputed by non-missing score used in previous visit. Analysis for change from baseline includes those with data available at baseline and visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 56
Units on a Scale | -2.3 (6.20)

2. Other Pre Specified Outcome: Change in the Crohn's Disease Activity Index (CDAI) Score From Baseline at Week 12
Description: The Crohn's Disease Activity Index is a composite score that is used to measure the clinical activity of Crohn's disease. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. Baseline was defined as the last non-missing record on or before the first dose of study drug.
Time Frame: Baseline to Week 12
Population: The ITT included all enrolled participants and received at least one dose of ozanimod. Analysis for change from baseline includes participants with data available at baseline and visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 54
Units on a Scale | -141.5 (99.42)

3. Other Pre Specified Outcome: Percentage of Participants With Clinical Remission Based on the Crohn's Disease Activity Index (CDAI) at Week 12
Description: Clinical Remission is defined as a CDAI score of < 150. The Crohn's Disease Activity Index is a composite score that is used to measure the clinical activity of Crohn's disease. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 12
Population: The ITT included all enrolled participants and received at least one dose of ozanimod. If CDAI score was missing, then non-responder imputation (NRI) was applied.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants | 33.3 [22.44 to 45.71]

4. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Clinical Response Based on Crohn's Disease Activity Index (CDAI) at Week 12
Description: Clinical Response is defined as a CDAI reduction from baseline of ≥ 100 points. The Crohn's Disease Activity Index is a composite score that is used to measure the clinical activity of Crohn's disease. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants | 50.7 [38.41 to 62.98]

5. Other Pre Specified Outcome: Percentage of Participants Who Achieved Clinical Remission Based on Patient-Reported Outcome (PRO2) Measure Definitions at Week 12
Description: The PRO2 is a composite score based on 2 components of the CDAI, the number of liquid or soft stools/day for 7 days, stool frequency (SF) and abdominal pain (AP) (rated on a scale of 0-3) assessed for 7 days. Clinical Remission (SF and AP remission) was defined as the average daily stool score ≤3 points AND average daily abdominal pain score ≤1 point. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 12
Population: The ITT included all enrolled participants and received at least one dose of ozanimod. If stool frequency and abdominal pain were missing, then non-reesponder imputation (NRI) was applied.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants | 20.3 [11.56 to 31.69]

6. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Clinical Response Based on Patient Reported Outcome (PRO2) Measures From Baseline at Week 12
Description: Clinical response based on PRO2 was defined as PRO2 decrease of ≥50% from baseline. The PRO2 is a composite score based on 2 components of the Crohn's Disease Activity Index, the number of liquid or soft stools/day for 7 days and the abdominal pain (rated on a scale of 0-3) assessed for 7 days. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 12
Population: The ITT included all enrolled participants and received at least one dose of ozanimod. If PRO2 CD score was missing, then non-responder imputation (NRI) was applied.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants | 29.0 [18.69 to 41.16]

7. Other Pre Specified Outcome: Percentage of Participants of Participants Who Achieved Endoscopic Remission Based on Simple Endoscopic Score for Crohn's Disease (SES-CD) Definitions at Week 12 (Paired Segments)
Description: Endoscopic remission is defined as SES-CD ≤ 4 points and a SES-CD decrease ≥ 2 points with no SES-CD sub-score >1point. The SES-CD assesses the degree of inflammation. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components are scored on a scale of 0 to 3. In the SES-CD, each of these 4 components are assessed in the five segments of the ileum and colon: ileum, right, transverse, left (descending and sigmoid), and rectum. The SES-CD is the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores is 0 - 12 for each segment, and 0 - 56 for the overall SES-CD score, with larger scores indicating greater severity of disease. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 12
Population: The ITT = all enrolled participants who received at least one dose of ozanimod. For paired segments analysis, any missing segment scores in the presence of at least 1 non-missing segmental SES-CD score were imputed by non-missing score used in the previous visit. If post-baseline SES-CD score was missing, then NRI was applied.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants | 10.1 [4.18 to 19.79]

8. Other Pre Specified Outcome: Percentage of Participants Who Achieved an Endoscopic Response-50 (Paired Segment) Based on Based on Simple Endoscopic Score for Crohn's Disease (SES-CD) Definitions at Week 12
Description: Endoscopic Response is defined as a SES-CD decrease from baseline of ≥ 50%. The SES-CD assesses the degree of inflammation. The SES-CD assesses the following 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components are scored on a scale of 0 to 3. In the SES-CD, each of these 4 components are assessed in the five segments of the ileum and colon: ileum, right, transverse, left (descending and sigmoid), and rectum. The SES-CD is the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores is 0 - 12 for each segment, and 0 - 56 for the overall SES-CD score, with larger scores indicating greater severity of disease. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 12
Population: The ITT included all enrolled participants and received at least one dose of ozanimod. For paired segments analysis, any missing segment scores in the presence of at least 1 non-missing segmental SES-CD score were imputed by non-missing score used in the previous visit. If post-baseline SES-CD score was missing, then NRI was applied.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants | 23.2 [13.87 to 34.91]

9. Other Pre Specified Outcome: Change in Roberts Intestinal Histopathology Index From Baseline (Paired Segments) at Week 12
Description: Changes in intestinal mucosa histopathologic features and disease activity were assessed by blinded pathologists. Robarts Histopathology Index (RHI) had a maximum total score of 165, with higher scores indicating more severe histological disease. Baseline was defined as the last non-missing record on or before the first dose of study drug.
Time Frame: Week 12
Population: The ITT population = all enrolled participants who received at least one dose of ozanimod. For paired segment analysis, any missing segment scores in the presence of at least 1 non-missing segmental SES-CD score were imputed by non-missing score used in the previous visit. Analysis includes participants with data available at baseline and visit.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 51
Units on a Scale | -10.2 (25.83)

10. Other Pre Specified Outcome: Improvement in Perianal and Enterocutaneous Fistulas
Description: The assessment is based on two parameters: whether the fistula is draining and whether it's open or closed. This is assessment was only on participants that had a fistula at baseline.
Time Frame: Week 12
Population: This endpoint was omitted because there were too few study participants with perianal or enterocutaneous fistulas at baseline to allow for meaningful evaluation. No analysis performed.
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Percentage of Participants Who Achieved Endoscopic Remission Based on Simple Endoscopic Score for Crohn's Disease (SES-CD) Definitions at Week 52 - Observed Cases
Description: as for outcome 7
Time Frame: Week 52
Population: The ITT = all enrolled participants who received at least one dose of ozanimod. For Robarts Observed Score, the SES-CD score was determined based on all available segments at a given visit without adjusting for the segments available at baseline. Observed Cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 30
Percentage of Participants | 16.7 [5.64 to 34.72]

12. Other Pre Specified Outcome: Percentage of Participants Who Achieved an Endoscopic Response-50 Based on Simple Endoscopic Score for Crohn's Disease (SES-CD) Definitions at Week 52
Description: as for outcome 8
Time Frame: Week 52
Population: The intent to treat population (ITT) = all enrolled participants who received at least one dose of ozanimod. For Robarts Observed Score, the SES-CD score is determined based on all available segments at a given visit without adjusting for the segments available at baseline.Observed cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 30
Percentage of Participants | 30.0 [14.73 to 49.40]

13. Other Pre Specified Outcome: Percentage of Participants Who Achieved Clinical Remission Based on the Crohn's Disease Activity Index (CDAI) at Week 52
Description: Clinical Remission is defined as a CDAI score of < 150. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 52
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. Observed Cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 32
Percentage of Participants | 65.6 [46.81 to 81.43]

14. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Clinical Response Based on CDAI at Week 52
Description: Clinical Response is defined as a CDAI reduction from baseline of ≥ 100 points. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 52
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. Observed Cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 32
Percentage of Participants | 93.8 [79.19 to 99.23]

15. Other Pre Specified Outcome: Percentage of Participants Who Achieved Clinical Remission Based on Patient-Reported Outcome (PRO2) Measure Definitions at Week 52
Description: Clinical Remission is defined as the participants with the average daily stool score ≤3 points AND average daily abdominal pain score ≤1 point. The PRO2 is a composite score based on 2 components of the CDAI, the number of liquid or soft stools/day for 7 days and the abdominal pain (rated on a scale of 0-3) assessed for 7 days.
Time Frame: Week 52
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. Observed cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 32
Percentage of Participants | 53.1 [34.74 to 70.91]

16. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Clinical Response Based on Patient Reported Outcome (PRO2) Measures From Baseline at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: The ITT included all enrolled participants and received at least one dose of ozanimod. Observed Cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 32
Percentage of Participants | 65.6 [46.81 to 81.43]

17. Other Pre Specified Outcome: Percentage of Participants in Clinical Remission Based on CDAI and PRO2 Definitions Who Were Off Corticosteroids at Week 52 of Those on Corticosteroids
Description: Clinical Remission is defined as CDAI score of < 150. The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease. The CDAI uses a questionnaire with responses scored numerically and weighted. The weighted sum of the 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, general well-being for 7 days, presence of complications, taking diarrhea medication, abdominal mass, hematocrit and percentage deviation from standard weight. The typical range of CDAI score is 0 to > 600. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Week 52
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. Participants who were taking corticosteroids at baseline. Observed cases.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 16
Percentage of Participants | 18.8 [4.05 to 45.65]

18. Other Pre Specified Outcome: Percentage of Participants With Clinical Remission Based on the Crohn's Disease Activity Index (CDAI) at Weeks 4 and 8
Description: Clinical Remission is defined as a CDAI score of < 150. The CDAI is a composite score that is used to measure the clinical activity of Crohn's disease. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Weeks 4 and 8
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. Non-responder imputed. (NRI).
Measure: Number; unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants
  Week 4 | 15.9
  Week 8 | 23.2

19. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Clinical Response Based on CDAI at Weeks 4 and 8
Description: Clinical Response is defined as a CDAI reduction from baseline of ≥ 100 points. The CDAI includes uses 8 components: Number of liquid or soft stools for 7 days, Abdominal pain for 7 days, General well-being for 7 days, Presence of complications, Taking diarrhea medication, Abdominal mass, Hematocrit and Percentage deviation from standard weight. Scores range from 0 to approximately 600, with higher scores indicating greater disease activity. 95% CI was created using the Clopper-Pearson Exact Method.
Time Frame: Weeks 4 and 8
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. If CDAI score was missing, then non-responder imputation was applied.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants
  Weeks 4 | 37.7
  Weeks 8 | 52.2

20. Other Pre Specified Outcome: Percentage of Participants Who Achieved Clinical Remission Based on Patient-Reported Outcome (PRO2) Measure Definitions at Weeks 4 and 8
Description: as for outcome 5
Time Frame: Weeks 4 and 8
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. If stool frequency and abdominal pain were missing, then non-reesponder imputation (NRI) was applied.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants
  Week 4 | 11.6
  Week 8 | 26.1

21. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Clinical Response Based on Patient Reported Outcome (PRO2) Measures at Weeks 4 and 8
Description: Clinical response based on PRO2 was defined as PRO2 decrease of ≥50%. The PRO2 is a composite score based on 2 components of the Crohn's Disease Activity Index, the number of liquid or soft stools/day for 7 days and the abdominal pain (rated on a scale of 0-3) assessed for 7 days. 95% confidence interval (CI) was created using the Clopper-Pearson Exact Method.
Time Frame: Weeks 4 and Week 8
Population: The ITT population included all enrolled participants who received at least one dose of ozanimod. If PRO2 CD score is missing, then Non-responder imputation (NRI) was applied.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of Participants
  Week 4 | 20.3
  Week 8 | 33.3

22. Other Pre Specified Outcome: Percentage of Participants With RHI Healing at Week 52
Description: Changes from baseline in intestinal mucosa histopathologic features and disease activity were assessed by blinded pathologists. Robarts Histopathology Index (RHI) had a maximum total score of 165, with higher scores indicating more severe histological disease. Baseline was defined as the last non-missing record on or before the first dose of study drug.
  The Robarts Histopathology Index (RHI) is a recently validated instrument that measures histological disease activity in ulcerative colitis.
  RHI Mucosal Healing was defined as a composite endpoint of being a responder for endoscopic remission and RHI remission.
Time Frame: Week 52
Population: The ITT population = all enrolled participants who received at least one dose of ozanimod. Observed cases.. Analysis includes participants with data available at baseline and visit.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 28
Percentage of Participants | 14.3 [4.03 to 32.67]

23. Other Pre Specified Outcome: Change in Fecal Calprotectin (Observed Cases) at Weeks 12 and 52
Description: Change in fecal calprotectin (observed cases) determined by comparing measurements at weeks 12 and 52 to baseline measurement.
Time Frame: Baseline to Weeks 12 and Week 52
Population: The intent to treat population (ITT) includes all enrolled participants who received at least one dose of ozanimod. Analysis for change from baseline includes participants with data available at baseline and visit.
Measure: Median (Full Range); unit: μg/g
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 46
μg/g
  Week 12 | -41.0 [-3518 to 4791]
  Week 52: number analyzed (Participants) | 31
  Week 52 | -103.3 [-4450 to 19534]

24. Other Pre Specified Outcome: Change in Serum C-Reactive Protein (CRP) Levels From Baseline (Observed Cases) at Weeks 12 and 52
Description: Change in Serum C-Reactive Protein was determined by comparing to baseline.
Time Frame: Baseline to Weeks 12 and 52
Population: as for outcome 23
Measure: Median (Full Range); unit: mg/L
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 53
mg/L
  Week 12 | 1.0 [-56 to 72]
  Week 52: number analyzed (Participants) | 32
  Week 52 | -0.5 [-59 to 41]

25. Other Pre Specified Outcome: Changes in Biomarkers: Percentage of Participants With CRP Response-10 - Non-responder Imputation
Description: The percentage of participants with a CRP Response-10 was assessed.
  CRP Response-10 is defined as C-reactive protein < 10 mg/L.
Time Frame: Week 12, Week 52
Population: The intent to treat population = all enrolled participants who received at least one dose of ozanimod.
  If any scores are missing then non-responder imputation is applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of participants
  Week 12 | 39.1 [27.60 to 51.63]
  Week 52 | 23.2 [13.87 to 34.91]

26. Other Pre Specified Outcome: Changes in Biomarkers: Percentage of Participants With FCP Response-250 - Non-responder Imputation
Description: The percentage of participants with a FCP Response-250 was assessed.
  FCP Response-250 is defined as Fecal calprotectin < 250 ug/g.
Time Frame: Week 12, Week 52
Population: The intent to treat population = all enrolled participants who received at least one dose of ozanimod.
  If any Fecal Calprotectin are missing then non-responder imputation is applied.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Percentage of participants
  Week 12 | 30.4 [19.92 to 42.69]
  Week 52 | 11.6 [5.14 to 21.57]

27. Other Pre Specified Outcome: Improvement in Perianal and Enterocutaneous Fistulas in Participants With Fistula's From Baseline at Weeks 4 and 8
Description: as for outcome 10
Time Frame: Baseline to Week 4 and 8
Population: as for outcome 10
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 0

28. Other Pre Specified Outcome: Pharmacokinetic Plasma Concentration of Ozanimod
Description: Summary of concentrations of Ozanimod in RPC01-2201 by scheduled visit.
Time Frame: From Day 1 to Week 52
Population: The intent to treat population = all enrolled participants who received at least one dose of ozanimod.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 66
pg/mL
  Day 1, post-dose | 48 (19)
  Week 4: number analyzed (Participants) | 63
  Week 4 | 228 (116)
  Week 8: number analyzed (Participants) | 59
  Week 8 | 195 (102)
  Week 12: number analyzed (Participants) | 56
  Week 12 | 165 (126)
  Week 24: number analyzed (Participants) | 43
  Week 24 | 190 (109)
  Week 52: number analyzed (Participants) | 33
  Week 52 | 154 (98)

29. Other Pre Specified Outcome: PK Plasma Concentration of Active Metabolite CC-112273
Description: Summary of concentrations of CC-112273 in RPC01-2201 by scheduled visit.
Time Frame: From Day 1 to Week 52
Population: The intent to treat population = all enrolled participants who received at least one dose of ozanimod.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 66
pg/mL
  Day 1, post-dose | 58 (41)
  Week 4: number analyzed (Participants) | 63
  Week 4 | 2348 (1289)
  Week 8: number analyzed (Participants) | 59
  Week 8 | 3138 (2129)
  Week 12: number analyzed (Participants) | 56
  Week 12 | 3507 (2337)
  Week 24: number analyzed (Participants) | 43
  Week 24 | 4259 (3322)
  Week 52: number analyzed (Participants) | 33
  Week 52 | 4055 (3569)

30. Other Pre Specified Outcome: Change From Baseline in Absolute Lymphocyte Count (ALC) Derived From Hematology Laboratory Results at Weeks 4, 8 and 12
Description: Change in Absolute Lymphocyte Count (ALC) from baseline was determined by comparied to baseline.
Time Frame: Baseline up to Weeks 4, 8 and 12
Population: The safety population included all enrolled participants who received at least one dose of ozanimod.
Measure: Mean (Standard Deviation); unit: 10 ^9 cells/L
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 65
10 ^9 cells/L
  Week 4: number analyzed (Participants) | 53
  Week 4 | -0.946 (0.783)
  Week 8: number analyzed (Participants) | 60
  Week 8 | -1.086 (0.778)
  Week 12: number analyzed (Participants) | 53
  Week 12 | -1.092 (0.783)

31. Secondary Outcome: The Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Induction and Extension Period
Description: A TEAE = any event with an onset date on or after the first dose date, or any ongoing event on the first dose date that worsens in severity or after the first dose date and until 90 days following the last dose of study drug treatment. An AE = untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product, which that does not necessarily have a causal relationship with the investigational treatment. An AE can be any unfavorable or unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product, whether or not considered related to the investigational medicinal product.
  A serious AE (experience) or reaction is any untoward medical occurrence that at any dose
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity, or
  * Is a congenital abnormality/birth defect
Time Frame: From the first day of ozanimod up to 90 days after the last dose of ozanimod; mean duration of exposure of study drug was 1.305 years
Population: The Safety population included all enrolled participants who received at least one dose of ozanimod.
Measure: Count of Participants; unit: Participants
Arm/Group | Ozanimod Hydrochloride (HCl) 1 mg
Number analyzed (Participants) | 69
Participants
  ≥ 1 TEAE | 59
  ≥ 1 Moderate or Severe TEAE | 43
  ≥ 1 Severe TEAE | 15
  ≥ 1 Possible, Probable or Related TEAE | 24
  ≥ 1 Related TEAE | 7
  ≥ 1 Serious TEAE | 18
  ≥ 1 Possible, Probable or Related Serious TEAE | 4
  ≥ 1 Related Serious TEAE | 1
  ≥ 1 TEAE Leading to Discontinuation of Ozanimod | 11
  ≥ 1 TEAE Leading to Study Withdrawal | 11
  Death | 1
  Death Possible, Probable or Related to Ozanimod | 1

ADVERSE EVENTS:
Time Frame: From the first day of ozanimod up to 90 days after the last dose of ozanimod; mean duration of exposure of study drug was 1.305 years
Groups:
- Ozanimod: Participants received ozanimod 1 mg capsules daily for the first 12 weeks of the induction period (an initial 7-day dose escalation regimen that consisted of 4 days of ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg) daily followed by 3 days of ozanimod HCl 0.5 mg (equivalent to ozanimod 0.46 mg) daily, with the final dose of ozanimod HCl 1 mg (equivalent to ozanimod 0.92 mg) daily dose reached on Day 8. Participants who completed the induction period had the opportunity at Week 12 to continue to receive ozanimod 1 mg capsules daily during the extension period up to an additional 148 weeks, provided that the investigator determined that the participant should continue. Participants in the extension period continued to receive ozanimod 1 mg capsules daily through Week 160. Participants who completed the Week 160 visit had the option to continue open-label ozanimod 1 mg capsules by immediately entering the open-label extension Phase 3 Crohn's Disease Study RPC01-3204.
Arm/Group | Ozanimod
All-Cause Mortality (participants affected / at risk) | 1/69
Serious Adverse Events (participants affected / at risk) | 18/69
Other Adverse Events (participants affected / at risk) | 47/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod (N=69)
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 6
Enterocolonic fistula (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Fistula of small intestine (Gastrointestinal disorders) | 1
Intestinal fistula (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Abdominal abscess (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal colic (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozanimod (N=69)
Anaemia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 10
Abdominal pain lower (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 6
Crohn's disease (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 5
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 5
C-reactive protein increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT02531113/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT02531113/SAP_001.pdf